CLINICAL TRIAL: NCT02254304
Title: Prospective Phase IV Clinical Trial on Effectiveness of Rebif Treatment of CIS and RMS Patients in Romania Using Electronic Device RebiSmart™
Brief Title: Effectiveness of Rebif® in Clinically Isolated Syndrome and Relapsing Multiple Sclerosis Using RebiSmart™
Acronym: PROCEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Romania SRL, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200136-583; 2014-001290-14 (EudraCT Number)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Relapsing Multiple Sclerosis; Clinically Isolated Syndrome
Keywords: Relapsing multiple sclerosis; Clinically isolated syndrome; RMS; CIS; RebiSmart™; Rebif®; Interferon beta-1a
MeSH Terms: interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rebif in Relapsing Multiple Sclerosis (RMS) Subjects (Experimental)
  Interventions: Drug: Rebif
- Rebif in Clinically Isolated Syndromes (CIS) Subjects (Experimental)
  Interventions: Drug: Rebif

INTERVENTIONS:
Drug: Rebif — Rebif will be administered at a dose of 44 microgram (mcg) subcutaneously using RebiSmart auto-injector three times a week for a total duration up to 12 months.
  Other Names: Interferon beta-1a

SUMMARY:
This is a Phase 4, interventional, multicenter study of subcutaneous Rebif® (interferon beta-1a) using RebiSmart™ device to assess effectiveness and adherence of treatment in subjects with clinically isolated syndrome (CIS) or relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between 18 to 65 years of age
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential as defined in the protocol
* Subjects diagnosed with CIS or RMS according to the revised McDonald criteria (2010)
* Treatment-naive subjects or subjects treated with Rebif® multi-dose injected by RebiSmart™ for no longer than 6 weeks prior to Baseline visit
* Subjects that are able to self-inject with RebiSmart™ (in the opinion of the physician)
* Subjects with Expanded Disability Status Scale (EDSS) score less than (<) 6 (inclusive) at Baseline
* Signed informed consent and subject data collection form

Exclusion Criteria:

* Subjects experiencing a relapse within 30 days before Baseline
* Participation in other studies within 30 days before Baseline
* Received any MS therapy within 6 months prior to study enrolment (for example, other disease-modifying drugs: immunomodulatory, immunosuppressive agents or combination therapy) with the exception of Rebif® multi-dose injected by RebiSmart™
* Any visual or physical impairment that precludes the subject from self-injecting the treatment using the RebiSmart™
* Pregnancy and breast-feeding
* Serious or acute heart disease such as uncontrolled cardiac dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure, as per investigator opinion
* Current or past (within the last 2 years) history of alcohol or drug abuse
* Have any contra-indications to treatment with interferon beta-1a according to Summary of Product Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please contact the Merck KGaA Communication Center, Darmstadt, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 sites in Romania.
Groups:
- Rebif In RMS Subjects: Rebif was administered in subjects with Relapsing Multiple Sclerosis (RMS) at a dose of 44 microgram (mcg) subcutaneously using RebiSmart auto-injector three times a week for a total duration up to 12 months.
- Rebif in CIS Subjects: Rebif was administered in subjects with Clinically Isolated Syndromes (CIS) at a dose of 44 microgram (mcg) subcutaneously using RebiSmart auto-injector three times a week for a total duration up to 12 months.
Period: Overall Study
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Started | 89 | 17
Completed | 75 | 13
Not Completed | 14 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Injection site pain and Injection fear | 1 | 0
Not completed — Personal causes | 4 | 1
Not completed — Personal decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects | Total
Number analyzed (Participants) | 89 | 17 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (10.71) | 31.6 (9.63) | 35.4 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 7 | 65
  Male | 31 | 10 | 41
Number of Subjects Living in City or Rural Area [Number; unit: subjects] — Number of subjects living in city or rural area were presented.
  subjects
    City | 71 | 13 | 84
    Rural | 18 | 4 | 22
Geographical Allocation [Number; unit: subjects] — Number of subjects depending upon the geographical location were presented.
  subjects
    North eastern | 18 | 3 | 21
    North western | 23 | 3 | 26
    South eastern | 45 | 10 | 55
    South western | 3 | 1 | 4
Nicotine Used Status [Number; unit: subjects] — Number of subjects with Nicotine used status was categorized under never used, regular user, occasional user and former user.
  subjects
    Never used | 63 | 10 | 73
    Regular user | 19 | 3 | 22
    Occasional user | 0 | 0 | 0
    Former user | 7 | 4 | 11
Alcohol Consumption [Number; unit: subjects]
  Subjects consumed alcohol | 3 | 1 | 4
  Subjects did not consume alcohol | 86 | 16 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Relapse-free RMS Subjects
Description: A relapse was defined as the appearance of a new symptom or worsening of an old symptom, attributable to multiple sclerosis (MS), accompanied by an appropriate new neurological abnormality or focal neurological dysfunction lasting at least 24 hours in the absence of fever, and preceded by stability or improvement for at least 30 days. Relapse-free RMS subjects were those who did not had relapse during 12 month treatment period. Data was planned to be reported for "Rebif in RMS Subjects" arm.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Rebif In RMS Subjects
Number analyzed (Participants) | 89
percentage of subjects | 66.3

2. Primary Outcome: Time to the First Relapse for CIS Subjects
Description: A relapse was defined as the appearance of a new symptom or worsening of an old symptom, attributable to MS, accompanied by an appropriate new neurological abnormality or focal neurological dysfunction lasting at least 24 hours in the absence of fever, and preceded by stability or improvement for at least 30 days. Time to the first relapse was defined as the duration from start of the treatment until first relapse. Data was planned to be reported for "Rebif in CIS Subjects" arm.
Time Frame: Baseline up to 12 months
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Rebif in CIS Subjects
Number analyzed (Participants) | 17
months | NA [NA to NA] — Median Kaplan Meier time to first relapse and inter-quartile range was not reached in the study because relapse was reported in only 1 subject.

3. Secondary Outcome: Percentage of Subjects With Treatment Adherence
Description: According to the World Health Organisation (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term). Percentage of subjects with treatment adherence under different categories (<=50%, >50-75%, >75-90%, >90%) were presented.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
percentage of subjects
  Adherence <=50% | 2.2 | 11.8
  Adherence >50-75% | 2.2 | 0.0
  Adherence >75-90% | 13.5 | 0.0
  Adherence >90% | 80.9 | 88.2
  Missing | 1.1 | 0.0

4. Secondary Outcome: Percentage of Subjects With Relapse by Adherence Category
Description: A relapse was defined as the appearance of a new symptom or worsening of an old symptom, attributable to multiple sclerosis (MS), accompanied by an appropriate new neurological abnormality or focal neurological dysfunction lasting at least 24 hours in the absence of fever, and preceded by stability or improvement for at least 30 days. According to the World Health Organisation (WHO), treatment adherence is defined as both compliance (taking the medication in the correct dose and according to the schedule prescribed) and persistency (maintenance of the drug regimen over the long-term). Percentage of subjects with relapses by adherence categories (<=50%, >50-75%, >75-90%, >90%) were presented. Adherence missing are the subjects who withdrew before 12 months and who did not have any relapses before withdrawal.
Time Frame: Month 12
Population: Full analysis set was used. Here "Number analyzed" signifies those subjects who were evaluable for specified categories. There were no subjects analyzed for certain categories (that is, "Number analyzed"= 0) because no subjects were evaluable for that arm in the specified category.
Measure: Number; unit: percentage of subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
percentage of subjects
  Relapse Status Yes, Adherence <= 50%: number analyzed (Participants) | 2 | 2
  Relapse Status Yes, Adherence <= 50% | 0.0 | 0.0
  Relapse Status Yes, Adherence >50-75%: number analyzed (Participants) | 2 | 0
  Relapse Status Yes, Adherence >50-75% | 0.0 |
  Relapse Status Yes, Adherence >75-90%: number analyzed (Participants) | 12 | 0
  Relapse Status Yes, Adherence >75-90% | 16.7 |
  Relapse Status Yes, Adherence >90%: number analyzed (Participants) | 72 | 15
  Relapse Status Yes, Adherence >90% | 19.4 | 6.7
  Relapse Status Yes, Adherence Missing: number analyzed (Participants) | 1 | 0
  Relapse Status Yes, Adherence Missing | 0.0 |
  Relapse Status No, Adherence <= 50%: number analyzed (Participants) | 2 | 2
  Relapse Status No, Adherence <= 50% | 0.0 | 50.0
  Relapse Status No, Adherence >50-75%: number analyzed (Participants) | 2 | 0
  Relapse Status No, Adherence >50-75% | 50.0 |
  Relapse Status No, Adherence >75-90%: number analyzed (Participants) | 12 | 0
  Relapse Status No, Adherence >75-90% | 50.0 |
  Relapse Status No, Adherence >90%: number analyzed (Participants) | 72 | 15
  Relapse Status No, Adherence >90% | 72.2 | 73.3
  Relapse Status No, Adherence Missing: number analyzed (Participants) | 1 | 0
  Relapse Status No, Adherence Missing | 0.0 |
  Relapse Status Missing, Adherence <=50%: number analyzed (Participants) | 2 | 2
  Relapse Status Missing, Adherence <=50% | 100.0 | 50.0
  Relapse Status Missing, Adherence >50-75%: number analyzed (Participants) | 2 | 0
  Relapse Status Missing, Adherence >50-75% | 50.0 |
  Relapse Status Missing, Adherence >75-90%: number analyzed (Participants) | 12 | 2
  Relapse Status Missing, Adherence >75-90% | 33.3 | 0.0
  Relapse Status Missing, Adherence >90%: number analyzed (Participants) | 72 | 15
  Relapse Status Missing, Adherence >90% | 8.3 | 20.0
  Relapse Status Missing, Adherence Missing: number analyzed (Participants) | 1 | 0
  Relapse Status Missing, Adherence Missing | 100.0 |

5. Secondary Outcome: Percentage of Subjects Who Prematurely Terminated Treatment and Reasons
Description: Percentage of subjects who prematurely terminated treatment and reasons were presented.
Time Frame: Baseline up to 12 months
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
percentage of subjects
  Adverse Event | 2.2 | 5.9
  Lost to follow-up | 2.2 | 11.8
  Protocol Non-compliance | 1.1 | 0.0
  Withdrew Consent | 3.4 | 0.0
  Pain at Injection site and fear of Injection | 1.1 | 0.0
  Personal causes | 4.5 | 5.9
  Personal decision | 1.1 | 0.0

6. Secondary Outcome: Percentage of Subjects Free From Clinical Disease Activity
Description: Expanded Disability Status Scale is abbreviated as EDSS.
Time Frame: Baseline up to 12 months
Population: Data could not be analyzed for this outcome because this is a composite outcome dependent on subjects free from relapses and EDSS progression, where EDSS progression requires to be collected every 3/6 months and confirmed 3/6 months later. Since EDSS progression was only done at Month 12, therefore this derived outcome could not be estimated.
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Subjects Free From Disability Progression
Description: Expanded Disability Status Scale is abbreviated as EDSS.
Time Frame: Baseline up to 12 months
Population: Data could not be analyzed for this outcome because this EDSS progression requires EDSS to be collected every 3/6 months and confirmed 3/6 months later. Since EDSS progression was only done at Month 12, therefore this derived outcome could not be estimated.
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean Number of Relapses in RMS Subjects
Description: A relapse was defined as the appearance of a new symptom or worsening of an old symptom, attributable to multiple sclerosis (MS), accompanied by an appropriate new neurological abnormality or focal neurological dysfunction lasting at least 24 hours in the absence of fever, and preceded by stability or improvement for at least 30 days.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: relapses
Arm/Group | Rebif In RMS Subjects
Number analyzed (Participants) | 89
relapses | 0.2 (0.54)

9. Secondary Outcome: Number of Subjects With Reasons of Missed Injections
Description: Number of subjects with the reasons of missed injections were presented. Aspartate transaminase and alanine transaminase are abbreviated as ALT and AST respectively. Glutamic oxaloacetic transaminase and glutamic pyruvic transaminase are abbreviated as GOT and GPT respectively.
Time Frame: Baseline up to 12 months
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment. Here "Number of Participants Analyzed" signifies number of subjects who missed the injections are evaluable for this outcome measure.
Measure: Number; unit: subjects
Groups:
- Rebif In RMS and CIS Subjects: Rebif was administered in RMS and CIS subjects at a dose of 44 mcg subcutaneously using RebiSmart auto-injector three times a week for a total duration up to 12 months.
Arm/Group | Rebif In RMS and CIS Subjects
Number analyzed (Participants) | 62
subjects
  Forgot to Injection | 48
  Tired | 23
  Fear of Injection | 11
  Did not want to have Injection | 5
  Pain at Injection site | 5
  Flu-like symptoms | 4
  Adverse event | 2
  Device broken | 1
  Device malfunctions | 1
  Device not functioning | 1
  Difficulty using the device | 1
  Elevated ALT and AST | 1
  Elevated liver enzymes | 2
  Increased GOT and GPT levels | 2
  Local erythema and induration | 1
  Missed study medication | 1
  Forgot the device at home | 1
  No access to medication | 1
  could not came at the scheduled visit | 1
  Patient redrawn intracutaneous | 1
  Stop the treatment | 1
  Technical problems with Rebismart | 1

10. Secondary Outcome: Overall Evaluation of RebiSmart Use as Assessed by Investigator
Description: Evaluation of RebiSmart was categorized under very easy, quite easy, Neither easy nor difficult, very difficult and missing
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
subjects
  Very easy | 46 | 13
  Quite easy | 32 | 1
  Neither easy nor difficult | 9 | 1
  Quite difficult | 0 | 0
  Very difficult | 1 | 2
  Missing | 1 | 0

11. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Visits to Clinic by Subjects Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of visits to clinic by subjects due to MS were presented.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment. Here "Number of Participants Analyzed" signifies number of subjects who visited clinic for MS.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
visits | 0.2 (0.49) | 0.1 (0.49)

12. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects Visiting Different Types of Doctors During Their Clinical Visit
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Subjects who took consultations with specialists, general practitioners for MS were presented.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment. Here "Number of Participants Analyzed" signifies number of subjects who visited to doctors for MS.
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 16 | 1
subjects
  General practitioner | 1 (0.49) | 1 (0.49)
  Specialist | 15 | 0

13. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Visits by Healthcare Professional to Subjects' Home
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of visits by healthcare professional to subjects' home were presented.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment. Here "Number of Participants Analyzed" signifies number of subjects evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
visits | 0.0 (0.11) | 0.0 (0.00)

14. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Times Subjects Visited Emergency Room Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of times subjects visited emergency room due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: emergency room visits
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
emergency room visits | 0.0 (0.00) | 0.0 (0.00)

15. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Days Subjects Hospitalized Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of days subjects hospitalized due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
days | 0.1 (0.75) | 0.0 (0.00)

16. Secondary Outcome: Healthcare Resource Utilization Questionnaire -Number of Subjects Who Paid Someone to Assist Them Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of subjects who paid someone to assist them due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
subjects | 2 (0.75) | 1 (0.00)

17. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Days Per Week Assistant Worked For Subject Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of days per week assistant worked for subject due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 2 | 1
days per week | 2.5 (2.12) | 2.0 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed.

18. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Hours Per Day Assistant Worked for Subject Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of hours per week assistant worked for subject due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 2 | 1
hours per day | 2.0 (1.41) | 4.0 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed.

19. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects Whose Relatives or Friends Missed Work Due to Subjects' Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of subjects whose relatives or friends missed work due to subjects' MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: subject
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
subject | 1 (1.41) | 1 (NA)

20. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Working Days Missed by Relative or Friend Due to Subjects' Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of working days missed by relative or friend due to subjects' MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 1 | 1
days | 1 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed. | 3 (NA) — Standard deviation could not be estimated as there was only 1 subject analyzed.

21. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects Who Missed Any Full Days From Work Due to Multiple Sclerosis (MS).
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of subjects who missed any full days from work due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
subjects | 2 (1.41) | 2 (NA)

22. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Full Days Missed From Work by Subjects
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of full days missed from work by subjects were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 2 | 2
days | 46.5 (61.52) | 3.5 (2.12)

23. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects Who Missed Any Partial Days From Work Due to Multiple Sclerosis (MS).
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of subjects who missed any partial days from work due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
subjects | 1 (1.41) | 2 (NA)

24. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Hours Per Day Missed From Work by Subjects
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of hours per day missed from work by subjects were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 1 | 2
hours per day | 8.0 (NA) — Standard deviation could not be estimated as there was only one subject analyzed. | 3.0 (2.83)

25. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects Accomplished Less Work Due to Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Number of subjects accomplished less work due to MS were presented.
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 88 | 17
subjects | 7 (NA) | 1 (2.83)

26. Secondary Outcome: Healthcare Resource Utilization Questionnaire - Number of Subjects With Percentage of Work Completed Despite of Multiple Sclerosis (MS)
Description: Subjects was assessed at Month 12 utilizing the Health Resource Utilization Questionnaire (HRUQ), a subject self-report tool designed to evaluate the economic impact of MS. Healthcare resource utilization was collected in the following areas: admissions and stays in the hospital, emergency room, consultations with specialists, general practitioners, or other healthcare professionals, work productivity, health care financial impact. Amount of work done by subjects in spite of multiple sclerosis was presented under different percentages (0-100%)
Time Frame: Month 12
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 7 | 1
Subjects
  0% Work Completed | 0 (NA) | 0 (2.83)
  10% Work Completed | 1 | 0
  20% Work Completed | 0 | 0
  30% Work Completed | 1 | 0
  40% Work Completed | 0 | 0
  50% Work Completed | 0 | 0
  60% Work Completed | 0 | 0
  70% Work Completed | 0 | 0
  80% Work Completed | 3 | 1
  90% Work Completed | 2 | 0
  100% Work Completed | 0 | 0

27. Secondary Outcome: Number of Subjects With Medication Adherence Based on Morisky Medication Adherence Score
Description: The Morisky Medication Adherence Scale (MMAS) is a valid and reliable instrument that consists of 8 items that measure medication adherence. The scores of the MMAS-8 range from 0 to 8. This self-report scale consists of 7 items answered with a yes or no and 1 item with a 5-point Likert scale. A score below 6 indicates low adherence, a score between 6 to < 8 indicates medium adherence and a score of 8 indicates high adherence.
Time Frame: Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: subjects
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
subjects
  Low Adherence | 23 | 3
  Medium Adherence | 45 | 6
  High Adherence | 21 | 8

28. Secondary Outcome: Number of Subjects With Adverse Event or Adverse Drug Reaction (AE/ADR), Serious AE/ADR, AE/ADR Leading to Death and AE/ADR Leading to Early Termination
Description: An AE was any untoward medical occurrence in a subject or clinical investigation in a subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An ADR was any unfavourable or unintended response (adverse event) that could possibly be related to drug treatment. An SAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. AE/ADR was planned to be reported for both the arms together.
Time Frame: Baseline up to 12 months
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Number; unit: subjects
Groups:
- Rebif: Rebif was administered in RMS and CIS subjects at a dose of 44 mcg subcutaneously using RebiSmart auto-injector three times a week for a total duration up to 12 months.
Arm/Group | Rebif
Number analyzed (Participants) | 106
subjects
  AE/ADR | 30
  Serious AE/ADR | 1
  AE/ADR Leading to Death | 0
  AE/ADR Leading to Early Termination | 4

29. Secondary Outcome: Expanded Disability Status Scale (EDSS) Score
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with MS. It consists of 8 ordinal rating scales assessing seven functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS).
Time Frame: Baseline, Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rebif In RMS Subjects | Rebif in CIS Subjects
Number analyzed (Participants) | 89 | 17
Units on a scale
  Baseline | 1.87 (0.991) | 1.24 (0.615)
  Month 12 | 1.80 (0.981) | 1.13 (0.581)

30. Secondary Outcome: Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: Baseline, Month 12
Population: Full analysis set included all subjects enrolled into the study and who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Kg/m^2
Arm/Group | Rebif In RMS and CIS Subjects
Number analyzed (Participants) | 106
Kg/m^2
  Baseline | 23.57 (3.347)
  Month 12 | 23.51 (3.582)

ADVERSE EVENTS:
Time Frame: Baseline up to 12 months
Description: AE/ADR was planned to be collected for both the arms together.
Arm/Group | Rebif
Serious Adverse Events (participants affected / at risk) | 1/106
Other Adverse Events (participants affected / at risk) | 15/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif (N=106)
Depression (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif (N=106)
Influenza Like Illness (General disorders) | 9
Hepatic Enzyme Increased (Investigations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other